CLINICAL TRIAL: NCT06891300
Title: Understanding and Treating Suicidal Ideation With Ketamine: A Diffusion Magnetic Resonance Imaging Study
Brief Title: Understanding and Treating Suicidal Ideation With Ketamine
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Royal's Institute of Mental Health Research (Other)
Responsible Party: Principal Investigator, Jennifer Phillips, Interim Scientific Director and Scientist, The Royal's Institute of Mental Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 0216; ECR-1-119-23 (Other Grant/Funding Number: American Foundation for Suicide Prevention (AFSP))
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideation; Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Suicidal Ideation; Ketamine; Neuroimaging
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): Participants will undergo a total of four IV ketamine infusions (0.5 mg/kg infused over 40 minutes), administered twice weekly for two weeks.
  Interventions: Drug: ketamine hydrochloride

INTERVENTIONS:
Drug: ketamine hydrochloride — Participants will undergo intravenous (IV) ketamine infusions (0.5 mg/kg infused over 40 minutes) under medical supervision. Treatments will be administered twice weekly for two weeks, for a total of four infusions.

SUMMARY:
The goal of this clinical trial is to treat active suicidal ideation in individuals with Major Depressive Disorder (MDD) using ketamine and to understand suicidal ideation by examining biological mechanisms using magnetic resonance imaging (MRI), and psychological mechanisms through validated clinical scales and qualitative interviews. The main questions it aims to answer are:

1. Will ketamine will reduce suicidal ideation in a significant proportion of study participants?
2. Will reduction in suicidal ideation will be accompanied by rapid changes in neuroimaging biomarkers?

Participants will receive four intravenous (IV) ketamine infusions administered twice weekly for two weeks. Participants will undergo two identical MRI scans: 1) within 48 hours prior to starting ketamine treatment, and 2) 24 hours after the fourth ketamine infusion. Suicidal ideation and depressive symptoms will be assessed prior to each imaging session alongside additional self-report measures. Qualitative interviews will occur within 72 hours after the fourth ketamine treatment.

DETAILED DESCRIPTION:
This innovative, mixed-method study will combine treatment, neuroimaging, and qualitative interview approaches in a clinical sample enriched for suicide-related outcomes and selected for the presence of active suicidal thoughts. For study participants, ketamine may offer a rapid strategy to alleviate suicidal ideation and provide a window of opportunity to engage in other, longer-term strategies to decrease suicide risk. Collecting longitudinal diffusion MRI data while patients undergo ketamine treatment will further the understanding of the key brain circuitry involved in suicidal ideation, and the mechanisms underlying ketamine's antisuicidal effects. This work may identify new targets for intervention and suicide prevention. Finally, seeking patient perspectives on their change in suicidal thinking with ketamine may allow them to gain insight into their own thought patterns and how they change with lessening of suicidal ideation. These unique findings have the potential to inform future research directions, provide support for existing theories of suicide, and may even lead to new theories.

The overarching goal of this project is to treat active suicidal ideation in patients with MDD using ketamine and to harness ketamine's rapid antisuicidal effects to understand suicidal ideation by examining biological mechanisms using MRI, and psychological mechanisms through validated clinical scales and qualitative interviews.

The central hypothesis is that ketamine will reduce suicidal ideation in a significant proportion of study participants and that reduction in suicidal ideation will be accompanied by rapid changes in neuroimaging biomarkers assessed using advanced diffusion MRI.

The specific aims of the study are to:

1. Measure changes in advanced diffusion MRI biomarkers (white matter microstructure, extracellular free water, and neurite density index) pre-post repeated ketamine treatment in association with changes in suicidal ideation.
2. Link changes in suicidal ideation pre-post ketamine treatment with changes in suicide-related psychological features including hopelessness, psychological pain, and perceived burdensomeness.
3. Explore patient perceptions of change in suicidal ideation while undergoing ketamine treatment through qualitative interviews.

This phase III, prospective, longitudinal study involves clinical assessment, neuroimaging, and qualitative interviews in participants undergoing repeated IV ketamine treatment for active suicidal ideation. The study is open-label and non-randomized. There is no use of a comparative agent. Participants will receive four IV ketamine infusions administered twice weekly for two weeks. Ketamine infusions will be administered at the BMO Innovative Clinic for Depression, a facility within the Royal Ottawa Mental Health Centre (ROMHC) that has safely administered over 500 intranasal esketamine treatments. Participants will undergo two identical MRI scans: 1) within 48 hours prior to starting treatment, and 2) 24 hours (+/-6 hours) after the fourth ketamine infusion. Suicidal ideation and depressive symptoms will be assessed prior to each imaging session alongside additional self-report measures. A short qualitative interview will occur within 72 hours after the fourth ketamine treatment. Each participants study duration is expected to be approximately 3 weeks total. The entire study will enroll participants over an 18 month period. Anticipated start date is MAR 2025 and anticipated end date is JAN 2026.

Thirty-six (36) participants will be recruited into the study. Systematic reviews and meta-analyses of the acute antisuicidal effects of ketamine report medium-large and large effect sizes. Despite calls for the reporting of standardized effect sizes in neuroimaging studies, existing preliminary diffusion MRI studies failed to report effect sizes for changes observed post-ketamine treatment. Nevertheless, assuming a medium effect size (Cohen's d=0.5), 80% power, a p value of 0.05, a power calculation shows a total sample size of 34 will allow detection of the primary outcome, pre-post treatment change in free water corrected fractional anisotropy. This sample size will inform future work. Early withdrawals will be replaced with new enrollments to allow 36 participants to complete the study.

The study team has extensive experience with longitudinal trials, and minimal attrition rate of participants is anticipated as the provision of treatment is expected to increase retention. Allowances have been made for participant withdrawal, incidental findings, or incomplete data by targeting a large enough sample size to inform future trials.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Ages 18-65 years old
3. Suicidal ideation severity score ≥3 on the Columbia Suicide Severity Rating Scale (C-SSRS) (Baseline/Screening version) at Screening Visit ("active suicidal ideation with any methods")
4. Diagnosis of Major Depressive Disorder (MDD) according to the Diagnostic and Statistical Manual for Mental Disorders 5th Edition (DSM-5)
5. Willing to maintain stable doses of concomitant medications throughout the study
6. Be under the care of a designated health care provider (i.e., family physician or psychiatrist) to follow their care after the completion of the study.

Exclusion Criteria:

1. Participants not medically cleared to receive ketamine treatment due to presence of clinically relevant disease (e.g., uncontrolled hypertension, renal or hepatic impairment, significant coronary artery disease, diabetes mellitus, seizure disorder).
2. Known or suspected hypersensitivity or intolerance to ketamine
3. Body mass index (BMI) ≥35
4. History of a primary psychotic disorder (e.g., schizophrenia), or current or recent (<2 years) acute episode of psychosis
5. Current and/or recent history (<12 months) of substance use/dependence (except for caffeine or nicotine) or problematic current alcohol use or dependence as defined by DSM-5 criteria
6. Pregnant, breastfeeding or of childbearing potential and unwilling to use an approved method of contraception during the study
7. History of significant head injury including loss of consciousness >5 minutes
8. Any MRI contraindications
9. Concurrent use of ketamine in any form
10. Concurrent active ECT or repetitive transcranial magnetic stimulation (rTMS) therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in white matter microstructure from pre-treatment to post-treatment, assessed via MRI. | Pre-treatment (up to -48 hours) to post-treatment (24+/-6 hours)
  Change in white matter microstructure (free water corrected fractional anisotropy) from pre-treatment to 24 hours post-treatment.

SECONDARY OUTCOMES:
Change in extracellular free water from pre-treatment to post-treatment, assessed via MRI. | Pre-treatment (up to -48 hours) to post-treatment (24+/-6 hours)
  Change in extracellular free water pre-post repeated ketamine infusions.
Change in neurite density index from pre-treatment to post-treatment, assessed via MRI. | Pre-treatment (up to -48 hours) to post-treatment (24+/-6 hours)
  Change in neurite density index pre-post repeated ketamine infusions.

OTHER OUTCOMES:
Change in suicidal ideation from pre-treatment to post-treatment, assessed via the Beck Suicide Scale (BSS). | Pre-treatment (up to -48 hours) to post-treatment (24+/-6 hours)
  Change in suicidal ideation from pre-treatment to post-treatment, as measured by the Beck Suicide Scale (BSS). The total BSS score can range from 0 to 38, with higher values indicating greater suicidal ideation severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Phillips, PhD, Principal Investigator — University of Ottawa Institute for Mental Health Research at The Royal
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD collected and stored within the Cardio-Neuro-Mind Data Platform (CNMDP) to which data sharing consent has been provided by the individual participant.